CLINICAL TRIAL: NCT03953300
Title: A Phase 4, Multicenter, Randomized, Double-blind, Parallel Group, Placebo Controlled Study to Evaluate the Effect of Benralizumab on Structural and Lung Function Changes in Severe Eosinophilic Asthmatics
Brief Title: Benralizumab Airway Remodeling Study in Severe Eosinophilic Asthmatics
Acronym: CHINOOK
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3250C00059; 2018-003391-13 (EudraCT Number)
Record Dates: First submitted 2019-04-10; First posted 2019-05-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Asthma
Keywords: Asthma; Eosinophilic Asthma; Lung Diseases; Inhaled Corticosteroids; ICS; LABA; benralizumab; Fasenra; mechanism of action; remodeling
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia; Lung Diseases | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Experimental): Administrated subcutaneously (SC) every 4 weeks for the first 3 doses, then every 8 weeks
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Administrated subcutaneously every 4 weeks for the first 3 doses, then every 8 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab: 30 mg/mL solution for injection in accessorized prefilled syringe (APFS) will be administered subcutaneously (SC) every 4 weeks for the first 3 doses - Weeks 0, 4 and 8, and then every 8 weeks - Weeks 16, 24, 32, 40.
  Arms: Benralizumab
Biological: Placebo — Matching placebo will be administered subcutaneously with accessorized prefilled syringe (APFS) every 4 weeks for the first 3 doses - Weeks 0, 4 and 8, and then every 8 weeks - Weeks 16, 24, 32, 40.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate effect of benralizumab on structural and lung function changes in severe eosinophilic asthmatics.

Changes will be assessed over 48 week treatment period in patients with persistent symptoms despite standard therapy of inhaled corticosteroids (ICS) plus long acting B2-agonist (LABA) with or without additional controller medication.

Patients who complete treatment will enter 4 weeks follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 through 70 years.
2. Physician-diagnosed asthma requiring continuous treatment with medium- or high-dose ICS plus LABA with or without additional controller medication for at least 12 months prior to Visit 1, and current treatment with high-dose ICS plus LABA for at least 3 months prior to Visit 1 with or without additional asthma maintenance medication.
3. Morning pre-BD FEV1 ≥50 to <80% of predicted normal value (PNV) and ≥1 liter (L) or morning pre-BD FEV1 ≥ 50 to < 90% of PNV, if historical pre-BD FEV1 value (within 12 months prior to screening visit) was < 80% of PNV.
4. A blood eosinophil count meeting any of 3 criteria: ≥300 cells/µL during screening or ≥ 220 to < 300 cells/μL during screening and documented eosinophil count of ≥ 300 cells/μL in the past 12 months, or ≥150 to <300 cells/µL during screening plus one of the following: presence of nasal polyps or pre-BD FVC <65% predicted at Visit 2
5. Negative pregnancy test.
6. Asthma control questionnaire (ACQ-6) >1.5.
7. Fewer than 12 exacerbations within the 6 months prior to Visit 3.

Exclusion Criteria:

1. Any disease or concomitant medication which could affect study results or safety of study participants, including:

   * current smokers
   * history of cancer
   * life-threatening asthma
   * clinically important pulmonary disease other than asthma
2. Use of chronic immunosuppressive medication or receipt of immunoglobulin (or blood products) within 30 days prior to the date informed consent is obtained.
3. Previously received:

   * benralizumab
   * live attenuated vaccines 30 days prior to the date of randomization.
   * bronchial thermoplasty in the last 24 months prior to Visit 1
   * any investigational non-biologic within 30 days (or 5 half-lives) prior to the date informed consent is obtained, whichever is longer.
   * any marketed or investigational biologic for the treatment of asthma within 4 months (or 5 half-lives) prior to the date informed consent is obtained, whichever is longer.
4. Currently pregnant, breastfeeding or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
The change in eosinophil numbers expressed as number/mm2 in submucosa as measured by major basic protein (MBP) staining in endobronchial biopsies | From baseline to Week 48 (Visit 10)
  The change in eosinophil numbers expressed as number/mm2 in submucosa as measured by major basic protein (MBP) staining in endobronchial biopsies
The change in airway wall area percentage as the overall median for airway generations 3 and 4 combined as measured by quantitative computed tomography (QCT) imaging | From baseline to Week 48 (Visit 10)
  The change in airway wall area percentage as the overall median for airway generations 3 and 4 combined as measured by quantitative computed tomography (QCT) imaging

SECONDARY OUTCOMES:
The change in eosinophil numbers, expressed as number/mm2 in epithelium as measured by major basic protein (MBP) staining in endobronchial biopsies | From baseline to Week 48 (Visit 10)
  The change in eosinophil numbers, expressed as number/mm2 in epithelium as measured by major basic protein (MBP) staining in endobronchial biopsies
The change in eosinophil numbers, expressed as number/mm2 in epithelium and submucosa as measured by major basic protein (MBP) staining in endobronchial biopsies | From baseline to Week 48 (Visit 10)
  The change in eosinophil numbers, expressed as number/mm2 in epithelium and submucosa as measured by major basic protein (MBP) staining in endobronchial biopsies
Absolute change in air trapping of the lung with expiratory density less than -856 Hounsfield Units (HU), and as expiratory-to-inspiratory ratio of mean lung density on computed tomography (CT) scans | From baseline to Week 48 (Visit 10)
  Absolute change in air trapping of the lung with expiratory density less than -856 Hounsfield Units (HU), and as expiratory-to-inspiratory ratio of mean lung density on computed tomography (CT) scans
Absolute change in air trapping/small airway obstruction derived from regional matching of the inspiratory/expiratory computed tomography (CT) scans | From baseline to Week 48 (Visit 10)
  Absolute change in air trapping/small airway obstruction derived from regional matching of the inspiratory/expiratory computed tomography (CT) scans
Change in airway lumen volume and airway resistance as measured by quantitative computed tomography (QCT) | From baseline to Week 48 (Visit 10)
  Change in airway lumen volume and airway resistance as measured by quantitative computed tomography (QCT)
Change in endobronchial biopsies on airway epithelial cell integrity | From baseline to Week 48 (Visit 10)
  Change in endobronchial biopsies on airway epithelial cell integrity
Change in endobronchial biopsies on reticular basement membrane (RBM) thickening | From baseline to Week 48 (Visit 10)
  Change in endobronchial biopsies on reticular basement membrane (RBM) thickening
Change in endobronchial biopsies on vascularization of the sub-mucosa | From baseline to Week 48 (Visit 10)
  Change in endobronchial biopsies on vascularization of the sub-mucosa
Assessments of peripheral airway resistance measured by AO | From baseline to Week 48 (Visit 10)
  Assessments of peripheral airway resistance measured by AO
Change in endobronchial biopsies on mucin 5AC, oligomeric mucus/gel-forming (MUC5AC) | From baseline to Week 48 (Visit 10)
  Change in endobronchial biopsies on mucin 5AC, oligomeric mucus/gel-forming (MUC5AC)
Absolute change in R5-R20 (peripheral airway resistance defined as the difference in resistance between 5 Hz [R5, total respiratory system resistance] and 20 Hz [R20, central resistance]) as measured by airwave oscillometry (AO) | From baseline to Week 48 (Visit 10)
  Absolute change in R5-R20 (peripheral airway resistance defined as the difference in resistance between 5 Hz [R5, total respiratory system resistance] and 20 Hz [R20, central resistance]) as measured by airwave oscillometry (AO)
Absolute change in area under the reactance curve (AX) as measured by airwave oscillometry (AO) | From baseline to Week 48 (Visit 10)
  Absolute change in area under the reactance curve (AX) as measured by airwave oscillometry (AO)
Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) residual volume (RV) | From baseline to Week 48 (Visit 10)
  Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) residual volume (RV)
Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) total lung capacity (TLC) | From baseline to Week 48 (Visit 10)
  Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) total lung capacity (TLC)
Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) inspiratory capacity (IC) | From baseline to Week 48 (Visit 10)
  Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) inspiratory capacity (IC)
Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) RV/TLC ratio | From baseline to Week 48 (Visit 10)
  Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) residual volume / total lung capacity (RV/TLC) ratio
Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP)functional residual capacity (FRC) | From baseline to Week 48 (Visit 10)
  Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP)functional residual capacity (FRC)
Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) vital capacity (VC) | From baseline to Week 48 (Visit 10)
  Absolute change in pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) vital capacity (VC)
Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP) residual volume (RV) | From baseline to Week 48 (Visit 10)
  Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP) residual volume (RV)
Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP) total lung capacity (TLC) | From baseline to Week 48 (Visit 10)
  Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP) total lung capacity (TLC)
Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP) inspiratory capacity (IC) | From baseline to Week 48 (Visit 10)
  Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP) inspiratory capacity (IC)
Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP) RV/TLC ratio | From baseline to Week 48 (Visit 10)
  Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP) residual volume / total lung capacity(RV/TLC) ratio
Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP)functional residual capacity (FRC) | From baseline to Week 48 (Visit 10)
  Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP)functional residual capacity (FRC)
Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP) vital capacity (VC) | From baseline to Week 48 (Visit 10)
  Absolute change in post-bronchodilator (BD) whole body plethysmogrpahy (WBP) vital capacity (VC)
Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP residual volume (RV) | From baseline to Week 48 (Visit 10)
  Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP residual volume (RV)
Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP total lung capacity (TLC) | From baseline to Week 48 (Visit 10)
  Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP total lung capacity (TLC)
Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP inspiratory capacity (IC) | From baseline to Week 48 (Visit 10)
  Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP inspiratory capacity (IC)
Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP RV/TLC ratio | From baseline to Week 48 (Visit 10)
  Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP residual volume / total lung capacity (RV/TLC) ratio
Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP functional residual capacity (FRC) | From baseline to Week 48 (Visit 10)
  Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP functional residual capacity (FRC)
Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP vital capacity (VC) | From baseline to Week 48 (Visit 10)
  Change from pre-bronchodilator (BD) whole body plethysmogrpahy (WBP) to post-BD WBP vital capacity (VC)
Change in post-bronchodilator (BD) forced expiratory volume in 1 second (FEV1) as measured by spirometry | From baseline to Week 48 (Visit 10)
  Change in post-bronchodilator (BD) forced expiratory volume in 1 second (FEV1) as measured by spirometry
Change in post-bronchodilator (BD) forced vital capacity (FVC) as measured by spirometry | From baseline to Week 48 (Visit 10)
  Change in post-bronchodilator (BD) forced vital capacity (FVC) as measured by spirometry
Change in post-bronchodilator (BD) FEV1/FVC as measured by spirometry | From baseline to Week 48 (Visit 10)
  Change in post-bronchodilator (BD) FEV1/FVC as measured by spirometry
Change in basophil number (number/mm2) in endobronchial biopsies as measured by immunohistochemistry (IHC) | From baseline to Week 48 (Visit 10)
  Change in basophil number (number/mm2) in endobronchial biopsies as measured by immunohistochemistry (IHC)
Absolute change from baseline to End of Treatment in mucus score assessed using computed tomography (CT) scans | From baseline to Week 48 (Visit 10)
  Absolute change from baseline to End of Treatment in mucus score assessed using computed tomography (CT) scans

OTHER OUTCOMES:
The number of Adverse events (AEs)/serious adverse events (SAEs). | From baseline to Week 52 (Visit 11)
  To evaluate the safety and tolerability of benralizumab. The number of Adverse events (AEs)/serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Mario Castro, MD, Principal Investigator — University of Kansas School of Medicine 3901 Rainbow Blvd. Kansas City, KS 66160, USA
Locations (35):
- United States (19):
  - Research Site, Birmingham, Alabama
  - Research Site, Los Angeles, California
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Snellville, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Ann Arbor, Michigan
  - Research Site, Bloomfield Hills, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Maspeth, New York
  - Research Site, New Bern, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Galveston, Texas
  - Research Site, Lewisville, Texas
  - Research Site, Mansfield, Texas
- Research Site, Calgary, Alberta, Canada
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Copenhagen
  - Research Site, Hvidovre
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Vejle
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Lund
- United Kingdom (6):
  - Research Site, Cambridge
  - Research Site, Headington
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Wythenshawe

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home